CLINICAL TRIAL: NCT04642898
Title: Increasing Treatment Efficacy Using SMART Methods for Personalizing Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shannon E. Sauer-Zavala (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Shannon E. Sauer-Zavala, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59307; R34MH123601-01 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Disorders; Post Traumatic Stress Disorder; Obsessive-Compulsive Disorder
Keywords: Unified Protocol; Cognitive Behavioral Therapy; Personalization
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Standard Group, Brief Intervention (Experimental): Participants in this group will receive 6 sessions of treatment in accordance with the standard, published Unified Protocol (UP) manual.
  Interventions: Behavioral: Standard UP Treatment
- Standard Group, Full Intervention (Experimental): Participants in this group will receive 12 sessions of treatment in accordance with the standard, published Unified Protocol (UP) manual.
  Interventions: Behavioral: Standard UP Treatment
- Capitalization Group, Brief Intervention (Experimental): Participants in this group will receive 6 sessions of treatment organized to prioritize skills that capitalize on patient strengths.
  Interventions: Behavioral: Capitalization UP Treatment
- Capitalization Group, Full Intervention (Experimental): Participants in this group will receive 12 sessions of treatment organized to prioritize skills that capitalize on patient strengths.
  Interventions: Behavioral: Capitalization UP Treatment
- Compensation Group, Brief Intervention (Experimental): Participants in this group will receive 6 sessions of treatment organized to prioritize skills that compensate for patient weaknesses.
  Interventions: Behavioral: Compensation UP Treatment
- Compensation Group, Full Intervention (Experimental): Participants in this group will receive 12 sessions of treatment organized to prioritize skills that compensate for patient weaknesses.
  Interventions: Behavioral: Compensation UP Treatment

INTERVENTIONS:
Behavioral: Standard UP Treatment — Participants will receive treatment modules sequenced in accordance with the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP; Barlow et al 2011; 2018).
  Arms: Standard Group, Brief Intervention; Standard Group, Full Intervention
Behavioral: Capitalization UP Treatment — Participants will receive Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) treatment modules organized to prioritize skills that capitalize on patient strengths.
  Arms: Capitalization Group, Brief Intervention; Capitalization Group, Full Intervention
Behavioral: Compensation UP Treatment — Participants will receive Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) treatment modules organized to prioritize skills that compensate for patient weaknesses.
  Arms: Compensation Group, Brief Intervention; Compensation Group, Full Intervention

SUMMARY:
The proposed study will determine the feasibility, tolerability, and acceptability of a study that tests: 1) personalized treatment delivery (i.e., module sequencing and treatment discontinuation timing) aimed at increasing the efficiency of care, and 2) the research protocol designed to evaluate the effects of this personalized care. A sample of 60 participants with heterogeneous anxiety disorders (and comorbid conditions, including depression) will be enrolled in a pilot sequential multiple assignment randomized trial (SMART). Patients will be randomly assigned to one of three sequencing conditions: transdiagnostic treatment administered in its standard module order, module sequences that prioritize capitalizing on relative strengths, and module sequences that prioritize compensating for relative weaknesses. Next, after 6 sessions, participants will be randomly assigned to either continue or discontinue treatment to evaluate post-treatment change at varying levels of target engagement. This proposal will enable us to 1) test the feasibility, acceptability, and tolerability of the research protocol, treatment sequencing conditions, and early treatment discontinuation, 2) determine whether a preliminary signal that capitalization or compensation module sequencing improves treatment efficiency exists, and 3) explore preliminary associations between core process engagement at treatment discontinuation and later symptom improvement. The proposed study, and the subsequent research it will support, will inform evidence-based decision rules to make existing treatments more efficient, ultimately reducing patient costs and increasing the mental health service system's capacity to address the needs of more individuals.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of at least one anxiety disorder, trauma- or stressor-related disorder, or obsessive-compulsive disorder
* fluent in English
* medication stability

Exclusion Criteria:

* concurrent therapy
* psychological condition that would be better addressed by alternative treatments
* have received more than 5 sessions of cognitive behavioral therapy in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sauer-Zavala, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Started | 11 | 10 | 10 | 10 | 10 | 10
Completed | 8 | 6 | 6 | 2 | 7 | 2
Not Completed | 3 | 4 | 4 | 8 | 3 | 8
Not completed — Withdrawal by Subject | 2 | 4 | 4 | 6 | 2 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Therapist left trial before patient completed treatment | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Ineligible due to conflict of interest with therapist | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant in the standard group, full intervention did not complete the demographic info survey and 1 participant in the compensation group, brief intervention did not report their age
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention | Total
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 10 | 10 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant in the standard group, full intervention did not complete the demographic info survey and 1 participant in the compensation group, brief intervention did not report their age
  years
    number analyzed (Participants) | 11 | 9 | 10 | 10 | 9 | 10 | 59
    (all) | 33.36 (8.87) | 39.67 (14.55) | 44.60 (15.10) | 36.10 (10.84) | 36.78 (10.84) | 37.50 (13.19) | 37.92 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant in the standard group, full intervention did not fill out the demographics form
  Participants
    number analyzed (Participants) | 11 | 9 | 10 | 10 | 10 | 10 | 60
    Female | 9 | 6 | 8 | 8 | 8 | 6 | 45
    Male | 2 | 3 | 2 | 2 | 2 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant in the standard group, full intervention did not fill out the demographics form
  Participants
    Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 2
    Not Hispanic or Latino | 10 | 9 | 10 | 9 | 10 | 10 | 58
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 0 | 1 | 3
  White | 9 | 7 | 10 | 9 | 9 | 9 | 53
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 10 | 10 | 10 | 10 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Severity From Baseline to 6 Weeks (Brief Intervention) or 12 Weeks (Full Intervention)
Description: Clinical severity will be measured using the Diagnostic Interview for Anxiety, Mood, and Obsessive Compulsive and Related Neuropsychiatric Disorders (DIAMOND) dimensional clinician ratings. Scores range from 1-7; higher scores indicate greater severity. Negative scores indicate symptom improvement.
Time Frame: Baseline to 6 weeks (Brief Intervention), Baseline to 12 weeks (Full Intervention
Population: Outcomes for participants in brief intervention groups will be the difference in clinical severity at assessments before and after 6 sessions of treatment. Outcomes for participants in full intervention groups will be the difference in clinical severity at assessments before and after 12 sessions of treatment. Participants who completed their pre- and post-treatment clinician assessment meetings were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Number analyzed (Participants) | 10 | 7 | 7 | 2 | 7 | 3
score on a scale | -2.40 (1.26) | -2.86 (1.46) | -2.71 (1.25) | -2.00 (1.14) | -3.00 (1.15) | -3.33 (.58)

2. Primary Outcome: Change in Self-Reported Anxiety Symptoms From Baseline to 6 Weeks (Brief Intervention) or 12 Weeks (Full Intervention)
Description: Anxiety symptoms will be measured using the Overall Anxiety Severity and Interference Scale (OASIS). This is a self-report measure in which scores range from 0-20; higher scores indicate more severe anxiety symptoms. Negative scores indicate symptom improvement. assessed at baseline and weekly for 6 or 12 weeks, change from baseline after 6 sessions (6 weeks) and after 12 sessions (12 weeks) are being reported
Time Frame: Baseline to 6 weeks (Brief Intervention), Baseline to 12 weeks (Full Intervention)
Population: Outcomes for participants in brief intervention groups is the difference in self-reported anxiety symptoms before and after 6 treatment sessions and outcomes for participants in full intervention groups is the difference in scores before and after 12 sessions. Participants who completed the pre- and post-treatment assessment questionnaires were analyzed. Several participants completed the post-treatment clinician meeting but not the questionnaires, creating a disparity in sample across outcomes
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Number analyzed (Participants) | 9 | 7 | 5 | 1 | 6 | 2
score on a scale | -2.56 (2.40) | -1.57 (4.69) | -2.00 (2.74) | -2.00 (0) | -3.33 (2.66) | -7.50 (.71)

3. Primary Outcome: Change in Self-Reported Depressive Symptoms From Baseline to 6 Weeks (Brief Intervention) or 12 Weeks (Full Intervention)
Description: Depressive symptoms will be measured using the Overall Depression Severity and Interference Scale (ODSIS). This is a self-report measure in which scores range from 0-20; higher scores indicate more severe anxiety symptoms. Negative scores indicate symptom improvement. assessed at baseline and weekly for 6 or 12 weeks, change from baseline after 6 sessions (6 weeks) and after 12 sessions (12 weeks) are being reported
Time Frame: Baseline to 6 weeks (Brief Intervention), Baseline to 12 weeks (Full Intervention)
Population: Outcomes for participants in brief intervention groups is the difference in self-reported symptoms before and after 6 treatment sessions and outcomes for participants in full intervention groups is the difference in scores before and after 12 sessions. Participants who completed the pre- and post-treatment assessment questionnaires were analyzed. Several participants completed the post-treatment clinician meeting but not the questionnaires, creating a disparity in sample across outcomes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Number analyzed (Participants) | 9 | 7 | 5 | 1 | 6 | 2
score on a scale | 0 (4.58) | -1.57 (6.32) | -1.20 (3.56) | -4.00 (0) | -1.67 (4.41) | -3.00 (1.41)

4. Primary Outcome: Change in Self-Reported Aversive Reactions to Emotions From Baseline to 6 Weeks (Brief Intervention) or 12 Weeks (Full Intervention)
Description: Aversive reactions to emotions will be measured using the distress aversion subscale of the Multidimensional Experiential Avoidance Questionnaire (MEAQ). This is a self-report measure in which scores range from 13-78; higher scores indicate greater negative reactions to emotional experiences. Negative scores indicate symptom improvement. assessed at baseline and weekly for 6 or 12 weeks, change from baseline after 6 sessions (6 weeks) and after 12 sessions (12 weeks) are being reported
Time Frame: Baseline to 6 weeks (Brief Intervention), Baseline to 12 weeks (Full Intervention)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Number analyzed (Participants) | 9 | 7 | 5 | 1 | 6 | 2
score on a scale | -4.44 (9.54) | -7.14 (6.79) | -3.40 (8.65) | -2.00 (0) | -6.83 (8.15) | -18.50 (6.36)

5. Primary Outcome: Change in Clinician-Rated Anxiety Symptoms From Baseline to 6 Weeks (Brief Intervention) or 12 Weeks (Full Intervention)
Description: Clinician-rated anxiety symptoms will be measured using the Hamilton Rating Scale for Anxiety Symptoms. Scores range from 0-56; higher scores indicate greater severity. Negative scores indicate symptom improvement. Outcomes for participants in brief intervention groups is the difference in clinician rated symptom scores before and after 6 treatment sessions and outcomes for participants in full intervention groups is the difference in clinician rated symptom scores before and after 12 sessions.
Time Frame: Baseline to 6 weeks (Brief Intervention), Baseline to 12 weeks (Full Intervention)
Population: Participants who completed the pre- and post-treatment clinician assessment meetings. Several participants completed the post-treatment clinician assessment, but did not complete the associated questionnaire batteries, which is why there is a disparity in the number of participants analyzed across outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Number analyzed (Participants) | 10 | 7 | 7 | 2 | 7 | 3
score on a scale | -3.6 (6.99) | -2.57 (7.5) | -8.29 (8.53) | -8.50 (7.78) | -6.00 (4.90) | -5.00 (8.19)

6. Primary Outcome: Change in Clinician-Rated Depressive Symptoms From Baseline to 6 Weeks (Brief Intervention) or 12 Weeks (Full Intervention)
Description: Clinician-rated depressive symptoms will be measured using the Hamilton Rating Scale for Depressive Symptoms. Scores range from 0-68; higher scores indicate greater severity. Negative scores indicate symptom improvement. Outcomes for participants in brief intervention groups is the difference in Clinician-Rated symptom scores before and after 6 treatment sessions and outcomes for participants in full intervention groups is the difference in Clinician-Rated symptom scores before and after 12 sessions.
Time Frame: Baseline to 6 weeks (Brief Intervention), Baseline to 12 weeks (Full Intervention)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
Number analyzed (Participants) | 9 | 7 | 7 | 2 | 7 | 3
score on a scale | -1.22 (3.77) | -.29 (7.15) | -6.86 (8.23) | -1.50 (3.54) | -3.86 (5.34) | -5.00 (3.46)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Standard Group, Brief Intervention | Standard Group, Full Intervention | Capitalization Group, Brief Intervention | Capitalization Group, Full Intervention | Compensation Group, Brief Intervention | Compensation Group, Full Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT04642898/Prot_SAP_ICF_001.pdf